CLINICAL TRIAL: NCT00440947
Title: See Detailed Description
Brief Title: Induction/Simplification With Atazanavir + Ritonavir + Abacavir/Lamivudine Fixed-Dose Combination In HIV-1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPZ108859
Record Dates: First submitted 2007-02-23; First posted 2007-02-27 (Estimated); Results first posted 2011-08-17 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2011-07

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: NORVIR; ARIES; EPZICOM; REYATAZ; HIV; simplification; Antiretroviral-naive
MeSH Terms: conditions — Infections; HIV Infections | interventions — abacavir; Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simplification (Other): Atazanavir (ATV) 400 mg QD + abacavir (ABC) 600 mg/lamivudine (3TC) 300 mg fixed dose combination (FDC) QD for 48 weeks followed by optional treatment extension for 60 weeks on the same regimen.
  Interventions: Drug: Abacavir (ABC)/lamivudine (3TC) + atazanavir (ATV)
- Continuation (Other): Atazanavir (ATV) 300 mg QD + ritonavir (/r) 100 mg QD + abacavir (ABC) 600mg/lamivuidine (3TC )300 mg FDC QD for 48 weeks followed by optional treatment extension for 60 weeks on the same regimen.
  Interventions: Drug: Abacavir (ABC)/lamivudine (3TC) + atazanavir (ATV) + ritonavir (/r)

INTERVENTIONS:
Drug: Abacavir (ABC)/lamivudine (3TC) + atazanavir (ATV) + ritonavir (/r) — Abacavir (ABC)/lamivudine (3TC) FDC + atazanavir (ATV)+ ritoanvir (/r) for 36weeks followed by ABC/3TC + ATV + /r for 48wks followed by optional treatment extension for 60 weeks on the same regimen
  Arms: Continuation
Drug: Abacavir (ABC)/lamivudine (3TC) + atazanavir (ATV) — Abacavir (ABC)/lamivudine (3TC) FDC + atazanavir (ATV) + ritonavir (/r) for 36 weeks followed by ABC/3TC + ATV for 48wks followed by optional treatment extension for 60 weeks on the same regimen
  Arms: Simplification

SUMMARY:
This study was designed to test the efficacy, safety, tolerability and durability of the antiviral response between atazanavir (ATV) + ritonavir (/r) + abacavir/lamivudine(ABC/3TC) Fixed dose combination (FDC) each administered once daily (QD) for 36 weeks followed by randomization to either a simplification regimen of ATV or continuation of ATV +/r for an additional 48 weeks, each in combination with ABC/3TC in antiretroviral (ART)-naive, HIV-1 infected, HLA-B*5701 negative subjects.

All subjects who complete the 84-week study will be eligible to enter the treatment extension phase and continue for an additional 60 weeks. The purpose of this extension is to obtain longer term treatment data in subjects who have completed the 84-week study.

DETAILED DESCRIPTION:
Safety and Efficacy of an Initial Regimen of Atazanavir (ATV) + Ritonavir (/r) + the Abacavir/Lamivudine Fixed-Dose Combination Tablet (ABC/3TC FDC) for 36 weeks followed by Simplification to Atazanavir with ABC/3TC FDC or Maintenance of the Initial Regimen for an Additional 48 weeks in Antiretroviral-Naive HIV-1 Infected HLA-B*5701 Negative Subjects followed by an Optional 60-Week Treatment Extension Phase

ELIGIBILITY:
Inclusion criteria:

* Subject is ≥ 18 years of age and has documented evidence of HIV-1 infection. (A female is eligible to enter and participate in this study if she is of: non child-bearing potential, child bearing potential with a negative pregnancy test and agrees to approved contraception methods, or agreement for complete abstinence.)
* Subject is antiretroviral-naïve (defined as having ≤14 days of prior therapy with any NRTI and no prior therapy with either a PI or NNRTI).
* Subject has plasma HIV-1 RNA ≥ 1,000 copies/mL by Roche COBAS AMPLICOR™ (Version 1.5) method at screening (if no other documentation of HIV infection is available, a positive result here may serve as documentation of HIV infection for this study).
* Subject is willing and able to understand and provide written informed consent prior to participation in this study.

Exclusion criteria:

* Subject is HLA-B*5701 positive.
* Subject testing positive for Hepatitis B or both Hepatitis B and Hepatitis C at screening (+ HbsAg)
* Genotyping results performed at the screening indicate that the subject has any of the following mutations at the reverse transcriptase (RT) enzyme: K65R, L74V, or Y115F, or a combination of two or more thymidine analog mutations (M41L, D67N, K70R, K219Q or E) that include changes at either L210 or T215, or ≥ 3 of the following protease mutations associated with atazanavir resistance: D30, V32, M36, M46, I47, G48, I50, I54, A71, G73, V77, V82, I84, N88, and L90.
* Women who are pregnant or breastfeeding.
* Subject has an active or acute CDC Clinical Category C event at screening. Treatment for the acute event must have been completed at least 30 days prior to screening.
* Subject is, in the opinion of the investigator, unable to complete the 84-week dosing period and protocol evaluations and assessments.
* Subject has ongoing clinically relevant pancreatitis or clinically relevant hepatitis at screening.
* Presence of a newly diagnosed HIV-related opportunistic infection or any medical condition requiring acute therapy at the time of enrollment.
* Subject suffers from a serious medical condition, such as diabetes, congestive heart failure, cardiomyopathy or other cardiac dysfunction (including known, clinically significant cardiac conduction system disease, severe first degree atrioventricular block [PR interval > 0.26 seconds], second or third-degree atrioventricular block), which in the opinion of the investigator would compromise the safety of the subject.
* Subject has pre-existing mental, physical, or substance abuse disorder, which in the opinion of the investigator would interfere with the subject's ability to comply with the dosing schedule and protocol evaluations and assessments.
* Subject has a history of inflammatory bowel disease or malignancy, intestinal ischemia, malabsorption, or other gastrointestinal dysfunction, which may interfere with drug absorption or render the subject unable to take oral medication.
* Subject requires treatment with foscarnet, hydroxyurea or other agents with documented activity against HIV-1 in vitro within 28 days of study administration.
* Subject requires treatment with immunomodulating agents (such as systemic corticosteroids, interleukins, vaccines, or interferons) within 28 days prior to screening, or subject had received an HIV-1 immunotherapeutic vaccine within 90 days prior to screening. Subjects using inhaled corticosteroids are eligible for enrollment.
* Creatinine clearance <50 mL/min via the Cockroft-Gault method [Cockroft, 1976].
* Active alcohol or substance use sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis or chemical hepatitis.
* Hypersensitivity to any component of the study drugs.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5 times the upper limit of normal (ULN).
* Total bilirubin > 1.5 times the upper limit of normal (ULN).
* Subject has any acute laboratory abnormality at screening, which, in the opinion of the investigator, would preclude the subject's participation in the study of an investigational compound. Any grade 4 laboratory abnormality would exclude a subject from study participation.
* Subject requires treatment with radiation therapy or cytotoxic chemotherapeutic agents within 28 days prior to screening, or has an anticipated need for these agents within the study period.
* Enrolled in one or more investigational drug protocols, which may have impacted HIV-1 RNA suppression.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
* Subjects requiring concomitant administration of proton pump inhibitors.
* Subjects who require treatment with the prohibited medications within 28 days of commencement of investigational product, or an anticipated need during the study.

Eligibility Criteria for Treatment Extension Phase:

-Subjects will be eligible to continue in the treatment extension phase (Weeks 84 to 144) if they have successfully completed the 84-week study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Actual)
Dates: Start 2007-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (50):
- United States (46):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Glastonbury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Ft. Pierce, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Somers Point, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greenville, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Norfolk, Virginia
- Canada (2):
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan

REFERENCES:
- [Background] L Ross, E Dejesus, M Potter, A LaMarca, D Murphy, I Melendez-Rivera, D Ward, P Wannamaker, J Uy, L Patel, H Amrine-Madsen, J Horton. Epidemiological and Genotypic Clustering of HIV infection within North America During 2007 International HIV & Hepatitis Drug Resistance Workshop & Curative Strategies, 8-12 June 2010, Dubrovnik, Croatia, Poster 150.
- [Background] Young B, Squires K, Patel P, Dejesus E, Bellos N, Berger D, Sutherland-Phillips DH, Liao Q, Shaefer M, Wannamaker P. First large, multicenter, open-label study utilizing HLA-B*5701 screening for abacavir hypersensitivity in North America. AIDS. 2008 Aug 20;22(13):1673-5. doi: 10.1097/QAD.0b013e32830719aa. PMID 18670229
- [Background] • L Ross, K Squires, B Young, E DeJesus, N Bellos, D Murphy, A Rachlis, H Zhao, L Patel, L Ross, P Wannamaker, M Shaefer. Genotypic Screening Impact in ARIES [Atazanavir (ATV) + Ritonavir (/r) + Abacavir/Lamivudine (ABC/3TC) for 36 Weeks Followed By Randomization to ATV +ABC/3TC or ATV/r + ABC/3TC for 48 Wks in HIV-infected, ART Naïve Patients] :Low Rates of Virologic Failure. The 19th Annual Canadian Conference on HIV/AIDS Research, 13-16 May 2010, Saskatoon, Canada. Poster P-169.
- [Background] K Squires, E DeJesus, N Bellos, D Ward, D Murphy, H Zhao, L Patel, L Ross, P Wannamaker, M Shaefer. Sustained Virologic Efficacy of Atazanavir (ATV) Versus Atazanavir/Ritonavir (ATV/r), each in Combination with Abacavir/Lamivudine (ABC/3TC) over 120 Weeks: the ARIES Trial. 48th ICAAC; September 12-15, 2010, Boston, MA. Poster H-204.
- [Background] K Squires, B Young, E DeJesus, N Bellos, D Murphy, D Sutherland-Phillips, H Zhao, L Patel, L Ross, P Wannamaker, M Shaefer. Atazanavir/Ritonavir (ATV/r) + Abacavir/Lamivudine (ABC/3TC) in Antiretroviral (ART)-Naive HIV-1 Infected HLA-B*5701 Negative Subjects Demonstrates Efficacy and Safety: the ARIES Trial. 48th ICAAC; October 25-28, 2008, Washington, DC. Poster H-1250a.
- [Background] K Squires, B Young, E DeJesus, N Bellos, D Murphy, D Sutherland-Phillips, H Zhao, L Patel, L Ross, P Wannamaker, M Shaefer. Similar Efficacy and Tolerability of Atazanavir (ATV) Compared to ATV/Ritonavir (RTV, r), Each in Combination with Abacavir/Lamivudine (ABC/3TC), after Initial Suppression with ABC/3TC + ATV/r in HIV-1 Infected Patients: 84 Week Results of the ARIES Trial. 5th IAS Conference; Cape Town, South Africa. Abstract WELBB103
- [Background] Squires KE, Young B, DeJesus E, Bellos N, Murphy D, Sutherland-Phillips DH, Zhao HH, Patel LG, Ross LL, Wannamaker PG, Shaefer MS; ARIES Study Team. Safety and efficacy of a 36-week induction regimen of abacavir/lamivudine and ritonavir-boosted atazanavir in HIV-infected patients. HIV Clin Trials. 2010 Mar-Apr;11(2):69-79. doi: 10.1310/hct1102-69. PMID 20542844
- [Background] Squires KE, Young B, Dejesus E, Bellos N, Murphy D, Zhao HH, Patel LG, Ross LL, Wannamaker PG, Shaefer MS; ARIES study team. Similar efficacy and tolerability of atazanavir compared with atazanavir/ritonavir, each with abacavir/lamivudine after initial suppression with abacavir/lamivudine plus ritonavir-boosted atazanavir in HIV-infected patients. AIDS. 2010 Aug 24;24(13):2019-27. doi: 10.1097/QAD.0b013e32833bee1b. PMID 20613461
- [Derived] Ross LL, Horton J, Hasan S, Brown JR, Murphy D, DeJesus E, Potter M, LaMarca A, Melendez-Rivera I, Ward D, Uy J, Shaefer MS. HIV-1 transmission patterns in antiretroviral therapy-naive, HIV-infected North Americans based on phylogenetic analysis by population level and ultra-deep DNA sequencing. PLoS One. 2014 Feb 26;9(2):e89611. doi: 10.1371/journal.pone.0089611. eCollection 2014. PMID 24586911
- [Derived] Squires KE, Young B, DeJesus E, Bellos N, Murphy D, Ward D, Zhao HH, Ross LL, Shaefer MS; ARIES Study Team. ARIES 144 week results: durable virologic suppression in HIV-infected patients simplified to unboosted atazanavir/abacavir/lamivudine. HIV Clin Trials. 2012 Sep-Oct;13(5):233-44. doi: 10.1310/hct1305-233. PMID 23134624
- [Derived] Young B, Squires KE, Ross LL, Santiago L, Sloan LM, Zhao HH, Wine BC, Pakes GE, Margolis DA, Shaefer MS; Aries EPZ108859 Study Team. Inflammatory biomarker changes and their correlation with Framingham cardiovascular risk and lipid changes in antiretroviral-naive HIV-infected patients treated for 144 weeks with abacavir/lamivudine/atazanavir with or without ritonavir in ARIES. AIDS Res Hum Retroviruses. 2013 Feb;29(2):350-8. doi: 10.1089/aid.2012.0278. Epub 2012 Dec 5. PMID 23039030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants (PAR) were recruited at 66 centers in the United States of America and Canada. HIV-RNA, human immunodeficiency virus-ribonucleic acid; ml, milliliters.
Pre-assignment Details: The study had a 36-week Non-randomized Induction Phase, followed by an 84-week Randomized Phase. All PAR completing 84 weeks were eligible to enter an optional 60-week extension phase (EP); some PAR chose not to continue in the EP. PAR whose HIV-RNA wasn't <50 copies/ml before Week 36 weren't allowed to randomize at Week 36 and were withdrawn.
Groups:
- ABC/3TC + ATV/r: Induction Phase: Abacavir (ABC) 600 milligrams (mg)/lamivudine (3TC) 300 mg fixed-dose combination tablet (FDC) once a day (QD) plus atazanavir (ATV) 300 mg QD + ritonavir (/r) 100 mg QD during the first 36 weeks of the study (planned interim analysis)
- ABC/3TC + ATV: Randomization Phase: Simplification regimen of the ABC/3TC FDC tablet administered QD for an additional 48 weeks in combination with 400 mg ATV QD
- ABC/3TC + ATV/r: Randomization Phase: Continuation of ABC/3TC FDC tablet administered QD for an additional 48 weeks in combination with ATV/r QD
- ABC/3TC + ATV: Extension Phase: Simplification regimen of the ABC/3TC FDC tablet administered QD for an additional 60 weeks in combination with ATV QD
- ABC/3TC + ATV/r: Extension Phase: Continuation of ABC/3TC FDC tablet administered QD for an additional 60 weeks in combination with ATV/r QD
Period: 36-Week Induction Phase
Arm/Group | ABC/3TC + ATV/r: Induction Phase | ABC/3TC + ATV: Randomization Phase | ABC/3TC + ATV/r: Randomization Phase | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Started | 515 | 0 | 0 | 0 | 0
Completed | 442 (23 PAR without confirmed HIV-RNA<50c/mL prior to Wk 36 couldn't be randomized but weren't withdrawn.) | 0 | 0 | 0 | 0
Not Completed | 73 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 16 | 0 | 0 | 0 | 0
Not completed — Insufficient Viral Load Response | 11 | 0 | 0 | 0 | 0
Not completed — Protocol-defined Virologic Failure | 5 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 10 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 16 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 7 | 0 | 0 | 0 | 0
Not completed — Kaposi Lesions Requiring Chemotherapy | 1 | 0 | 0 | 0 | 0
Not completed — Took Exclusionary Medications | 1 | 0 | 0 | 0 | 0
Not completed — Genotype Had Exclusionary Mutations | 1 | 0 | 0 | 0 | 0
Not completed — Fleeing Police; Outstanding Warrants | 1 | 0 | 0 | 0 | 0
Not completed — Incarceration | 3 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Period: 48-Week Randomization Phase
Arm/Group | ABC/3TC + ATV/r: Induction Phase | ABC/3TC + ATV: Randomization Phase | ABC/3TC + ATV/r: Randomization Phase | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Started | 0 | 210 | 209 | 0 | 0
Completed | 0 | 194 | 185 | 0 | 0
Not Completed | 0 | 16 | 24 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 5 | 0 | 0
Not completed — Protocol-defined Virologic Failure | 0 | 1 | 1 | 0 | 0
Not completed — Non-compliance | 0 | 3 | 4 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 8 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 4 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0
Not completed — Incarceration | 0 | 3 | 0 | 0 | 0
Not completed — Trying to Get Pregnant | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 2 | 0 | 0 | 0
Period: Optional 60-Week Extension Phase
Arm/Group | ABC/3TC + ATV/r: Induction Phase | ABC/3TC + ATV: Randomization Phase | ABC/3TC + ATV/r: Randomization Phase | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Started | 0 | 0 | 0 | 189 | 180
Completed | 0 | 0 | 0 | 160 | 154
Not Completed | 0 | 0 | 0 | 29 | 26
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 3
Not completed — Insufficient Viral Load Response | 0 | 0 | 0 | 1 | 1
Not completed — Protocol-defined Virologic Failure | 0 | 0 | 0 | 3 | 2
Not completed — Non-compliance | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9 | 9
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 3
Not completed — Pregnancy | 0 | 0 | 0 | 3 | 0
Not completed — Participant Moved | 0 | 0 | 0 | 1 | 1
Not completed — Sponsor Request | 0 | 0 | 0 | 1 | 1
Not completed — Sponsor Terminated Site | 0 | 0 | 0 | 3 | 3
Not completed — Other | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Participant Remained in Cuba | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ABC/3TC + ATV/r: All participants starting the Induction Phase: ABC 600 mg/3TC 300 mg FDC tablet QD plus ATV 300 mg QD + /r 100 mg QD during the first 36 weeks of the study (planned interim analysis)
Arm/Group | ABC/3TC + ATV/r
Number analyzed (Participants) | 515
Age Continuous [Mean (Standard Deviation); unit: Years] | 38.3 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 429
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 167
  American Indian or Alaskan Native | 9
  Asian - Central/South Asian Heritage | 4
  Asian - East Asian Heritage | 3
  Asian - Japanese Heritage | 1
  Asian - South East Asian Heritage | 3
  Native Hawaiian or Other Pacific Islander | 1
  White - Arabic/North African Heritage | 5
  White - White/Caucasian/European Heritage | 316
  Mixed Race | 6
Number of participants with the indicated baseline HIV-RNA level [Number; unit: participants] — HIV-1 RNA, Human Immunodeficiency Virus type 1 Ribonucleic acid. HIV-1 viral load was measured as virus copies per milliliter (ml) at baseline.
  participants
    HIV-1 RNA <100,000 | 227
    HIV-1 RNA 100,000-<250,000 | 143
    HIV-1 RNA 250,000-<500,000 | 73
    HIV-1 RNA >=500,000 | 72
Number of participants with the indicated Baseline CD4+ Cell Count [Number; unit: participants] — A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts.
  participants
    CD4+ cells <50 | 69
    CD4+ cells 50-<200 | 190
    CD4+ cells >=200 | 256
Number of participants with the indicated Center for Disease Control (CDC) Classification [Number; unit: participants] — AIDS, Acquired Immunodeficiency Syndrome CDC classifications are Asymptomatic, Symptomatic, or AIDs.
  participants
    Asymptomatic HIV Infection | 353
    Symptomatic (non-AIDS) condition | 97
    AIDS | 65
Median Baseline CD4+ Cell Count [Median (Full Range); unit: cells per cubic millimeter] | 199 [19 to 754]
Median Baseline HIV-1 RNA Level [Median (Full Range); unit: log10 copies/ml] | 5.076 [2.989 to 6.620]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants (PAR) Who Achieved Plasma HIV-1 RNA <50 Copies (c) /Milliliter (ml) at the Week 84 Visit
Description: The percentage of PAR with HIV-1 RNA virus <50 c/ml determined from a blood sample drawn at Week 84 was tabulated by treatment arm with stratification by baseline HIV-1 RNA (<100,000 c/ml and >=100,000 c/ml). Per TLOVR algorithm, responders were PAR with confirmed viral load <50 c/ml who had not met any non-responder criterion. Non-responders were PAR who never achieved confirmed HIV RNA <50 c/ml, prematurely discontinued study or study medication for any reason, had confirmed rebound to at least 50 c/ml, or had an unconfirmed HIV RNA of at least 50 c/ml at last visit.
Time Frame: Week 84
Population: Intent-to-Treat (ITT)-Exposed Population, Randomized Phase: all PAR exposed to at least one dose of study medication during the Randomized Phase of the study. The primary analysis method was time to loss of virologic response (TLOVR) for the proportion of PAR with HIV-1 RNA <50 c/ml at Week 84 in the Simplification arm and Continuation arms
Measure: Number; unit: percentage of participants
Groups:
- ABC/3TC + ATV: Randomized Phase: Randomized Phase: simplification regimen of the ABC/3TC FDC tablet administered QD for an additional 48 weeks in combination with ATV QD
- ABC/3TC + ATV/r: Randomized Phase: Randomized Phase: continuation of ABC/3TC FDC tablet administered QD for an additional 48 weeks in combination with ATV/r QD
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 210 | 209
percentage of participants | 86 | 81
Statistical Analysis 1: Comparison: ABC/3TC + ATV: Randomized Phase vs ABC/3TC + ATV/r: Randomized Phase; Test type: Non-Inferiority or Equivalence — Non-inferiority would be established between the two arms if the lower limit of the 2-sided 95% confidence interval (CI) on the difference in the percentage of participants with HIV-1 RNA <50 c/mL at Week 84 was -12% or greater; p = 0.140, Cochran-Mantel-Haenszel; p-value was obtained from Cochran-Mantel-Haenszel stratified by baseline HIV-1 RNA (<100000/>=100000); Risk Difference (RD) = 5.4, 95% CI 2-sided [-1.8 to 12.5]

2. Secondary Outcome: Mean Age at Baseline of Participants Randomized to Treatment for the 48-Week Randomized Phase
Description: The mean age of participants randomized to treatment in the Randomized Phase was calculated at Baseline.
Time Frame: Baseline of Randomized Phase
Population: ITT-E Population: all participants exposed to at least one dose of study medication during the Randomized Simplification Phase
Measure: Mean (Standard Deviation); unit: years
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 210 | 209
years | 37.5 (10.23) | 39.7 (9.71)

3. Secondary Outcome: Percentage of Participants Who Achieved Plasma HIV-1 RNA <50 c/ml at the Week 36 Visit
Description: The percentage of PAR with HIV-1 RNA virus <50 c/ml from a Week 36 blood sample was tabulated. Per TLOVR algorithm, responders were PAR with confirmed viral load <50 c/ml who had not met any non-responder criterion. Non-responders were PAR who never achieved confirmed HIV RNA <50 c/ml, prematurely discontinued (DC) study or study medication (any reason), had confirmed rebound to >=50 c/ml, or had an unconfirmed HIV RNA >=50 c/ml at last visit. ITT-E observed analysis (Obs): all observed data. ITT-E M/D=F analysis: PAR with missing data/data collected after study medication DC were failures.
Time Frame: Week 36
Population: ITT-E Population, Induction Phase: all participants exposed to at least one dose of study medication during the Induction Phase of the study
Measure: Number; unit: percentage of participants
Groups:
- ABC/3TC + ATV/r: Induction Phase: Induction Phase: ABC 600 mg/3TC 300 mg FDC tablet QD plus ATV 300 mg QD + /r 100 mg QD during the first 36 weeks of the study (planned interim analysis)
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 515
percentage of participants
  TLOVR | 80
  Obs | 88
  M/D=F | 77

4. Secondary Outcome: Percentage of Participants Who Achieved Plasma HIV-1 RNA <50 c/ml at the Week 84 Visit
Description: A blood sample was drawn to determine the amount of HIV-1 RNA virus in c/ml at Week 84. The percentage of participants with HIV-1 RNA <50 c/ml at Week 84 was tabulated. The secondary analysis methods were: Observed (Obs; uses all visits with data in the analysis period), and missing/discontinuation=failure (M/D=F) analyses. M/D=F: participants with missing data or data collected after study medication DC were considered failures.
Time Frame: Week 84
Population: ITT-E Population, Randomized Phase. The secondary analysis methods were Observed (Obs) and missing/discontinuation=failure (M/D=F) analyses.
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 210 | 209
percentage of participants
  Obs | 92 | 92
  M/D=F | 85 | 82

5. Secondary Outcome: Percentage of Participants Who Achieved Plasma HIV-1 RNA <50 c/ml at the Week 144 Visit
Description: Percentage of PAR with HIV-1 RNA <50 c/ml at Week 144 was tabulated; stratified by baseline HIV-1 RNA (<100,000 and >=100,000 c/ml). Per TLOVR algorithm, responders were PAR with confirmed (CF) HIV RNA <50 c/ml who had not met any non-responder (NR) criterion. NR were PAR who never achieved CF HIV RNA <50 c/ml, prematurely discontinued (DC) study or study medication (Med), had CF rebound to >=50 c/ml, or had an unconfirmed HIV RNA >=50 c/ml at last visit. Observed analysis (Obs): all observed data. M/D=F analysis: PAR with missing data/data collected after study Med DC were failures.
Time Frame: Week 144
Population: ITT-Extension Population, Extension Phase: all participants exposed to at least one dose of study medication during the Extension Phase of the study
Measure: Number; unit: percentage of participants
Groups:
- ABC/3TC + ATV: Extension Phase: Extension Phase: simplification regimen of the ABC/3TC FDC tablet administered QD for an additional 60 weeks in combination with ATV QD
- ABC/3TC + ATV/r: Extension Phase: Extension Phase: continuation of ABC/3TC FDC tablet administered QD for an additional 60 weeks in combination with ATV/r QD
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 189 | 180
percentage of participants
  TLOVR | 77 | 73
  Obs | 95 | 92
  M/D=F | 80 | 78

6. Secondary Outcome: Percentage of Participants Who Achieved Plasma HIV-1 RNA <400 c/ml at the Week 36 Visit
Description: The percentage of PAR with HIV-1 RNA virus <400 c/ml from a Week 36 blood sample was tabulated. Per TLOVR algorithm, responders were PAR with confirmed (CF) HIV RNA <400 c/ml who had not met any non-responder criterion. Non-responders were PAR who never achieved CF HIV RNA <400 c/ml, prematurely discontinued (DC) study or study medication (Med; any reason), had CF rebound to >=400 c/ml, or had an unconfirmed HIV RNA >=400 c/ml at last visit. ITT-E observed analysis (Obs): all observed data. ITT-E M/D=F analysis: PAR with missing data/data collected after study Med DC were failures.
Time Frame: Week 36
Population: ITT-E Population, Induction Phase
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 515
percentage of participants
  TLOVR | 82
  Obs | 98
  M/D=F | 84

7. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA <400 c/ml at the Week 84 Visit
Description: Percentage of PAR with HIV-1 RNA <400 c/ml at Week 84 was tabulated; stratified by baseline HIV-1 RNA (<100,000 and >=100,000 c/ml). Per TLOVR algorithm, responders were PAR with confirmed (CF) HIV-RNA <400 c/ml who had not met any non-responder (NR) criterion. NR were PAR who never achieved CF HIV RNA <400 c/ml, prematurely discontinued (DC) study or study medication (Med), had CF rebound to >=400 c/ml, or had an unconfirmed HIV RNA >=400 c/ml at last visit. Observed analysis (Obs): all observed data. M/D=F analysis: PAR with missing data/data collected after study Med DC were failures.
Time Frame: Week 84
Population: ITT-E Population, Randomized Phase
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 210 | 209
percentage of participants
  TLOVR | 92 | 86
  Obs | 99 | 98
  M/D=F | 92 | 87

8. Secondary Outcome: Percentage of Participants Who Achieved HIV-1 RNA <400 c/ml at the Week 144 Visit
Description: Percentage of PAR with HIV-1 RNA <400 c/ml at Week 144 was tabulated; stratified by baseline HIV-1 RNA (<100,000 and >=100,000 c/ml). Per TLOVR algorithm, responders were PAR with confirmed (CF) HIV-RNA <400 c/ml who had not met any non-responder (NR) criterion. NR were PAR who never achieved CF HIV RNA <400 c/ml, prematurely discontinued (DC) study or study medication (Med), had CF rebound to >=400 c/ml, or had an unconfirmed HIV RNA >=400 c/ml at last visit. Observed analysis (Obs): all observed data. M/D=F analysis: PAR with missing data/data collected after study Med DC were failures.
Time Frame: Week 144
Population: ITT-Extension Population, Extension Phase
Measure: Number; unit: percentage of participants
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 189 | 180
percentage of participants
  TLOVR | 84 | 80
  Obs | 99 | 97
  M/D=F | 84 | 82

9. Secondary Outcome: Number of Participants Who Met the Protocol-defined Virologic Failure (PDVF) Criteria at Week 36
Description: The number of participants that failed to respond to therapy through 36 weeks on treatment, based on the protocol definition of virologic failure (PDVF), was tabulated. PDVF was defined as (a) failure to achieve plasma HIV-1 RNA <400 c/ml by Week 30 or (b) confirmed HIV-1 RNA rebound >=400 c/ml after achieving HIV-1 <400 c/ml.
Time Frame: Week 36
Population: ITT-E Population, Induction Phase
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 515
participants
  Protocol-defined virologic failure | 15
  Failure to achieve <400 c/ml by Week 30 | 5
  Confirmed rebound after achieving <400 c/ml | 10

10. Secondary Outcome: Number of Participants Who Met the PDVF Criteria at Week 84
Description: The number of participants that failed to respond to therapy from the time of treatment randomization through Week 84, based on the protocol definition of virologic failure (PDVF), was tabulated. PDVF was defined as (a) failure to achieve plasma HIV-1 RNA <400 c/ml by Week 30 or (b) confirmed HIV-1 RNA rebound >=400 c/ml after achieving HIV-1 <400 c/ml.
Time Frame: Week 84
Population: ITT-Exposed Population, Randomized Phase. TLOVR. One participant met PDVF criteria at Week 36 and was included in the Week 36 PDVF but had been randomized; this participant is therefore also included in this PDVF tabulation.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 210 | 209
participants
  Protocol-defined virologic failure | 1 | 7
  Confirmed rebound after achieving <400 c/ml | 1 | 7

11. Secondary Outcome: Number of Participants Who Met the PDVF Criteria at Week 144
Description: The number of participants enrolled in the extension phase that failed to respond to therapy from Week 84 through Week 144, based on the protocol definition of virologic failure (PDVF) was tabulated,. PDVF was defined as (a) failure to achieve plasma HIV-1 RNA <400 c/ml by Week 30 or (b) confirmed HIV-1 RNA rebound >=400 c/ml after achieving HIV-1 <400 c/ml.
Time Frame: Week 144
Population: ITT-Extension Population, Extension Phase. TLOVR.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 210 | 209
participants
  Protocol-defined virologic failure | 5 | 6
  Confirmed rebound after achieving <400 c/ml | 5 | 6

12. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 36
Description: Change from baseline was calculated as the Week 36 value minus the baseline value. Blood was drawn to analyze for plasma HIV viral load.
Time Frame: Baseline and Week 36
Population: ITT-E Population, Induction Phase. Observed Population. Participants could only be included in the analysis if they had completed a Week 36 visit and had a viral load result obtained during that visit period.
Measure: Mean (Standard Deviation); unit: log10 c/ml
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 447
log10 c/ml | -3.241 (0.775)

13. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 84
Description: Change from baseline was calculated as the Week 84 value minus the baseline value. Blood was drawn to analyze for plasma HIV viral load.
Time Frame: Baseline and Week 84
Population: ITT-E Population, Randomized Phase. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 84 visit and had a viral load result obtained during that visit period.
Measure: Mean (Standard Deviation); unit: log10 c/ml
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 194 | 187
log10 c/ml | -3.261 (0.681) | -3.270 (0.698)

14. Secondary Outcome: Change From Baseline in HIV-1 RNA at Week 144
Description: Change from baseline was calculated as the Week 144 value minus the baseline value. Blood was drawn to analyze for plasma HIV viral load.
Time Frame: Baseline and Week 144
Population: ITT-Extension Population, Extension Phase. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 144 visit and had a viral load result obtained during that visit period.
Measure: Mean (Standard Deviation); unit: log10 c/ml
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 163 | 154
log10 c/ml | -3.291 (0.675) | -3.239 (0.835)

15. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 36
Description: Blood was drawn to analyze for CD4+ cell count. A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts. Change from baseline was calculated as the Week 36 value minus the baseline value.
Time Frame: Baseline and Week 36
Population: ITT-E Population, Induction Phase. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 36 visit and had a cell count obtained during that visit period.
Measure: Mean (Standard Deviation); unit: cells/millimeters cubed (mm^3)
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 438
cells/millimeters cubed (mm^3) | 185.4 (121.84)

16. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 84
Description: A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts. Change from baseline was calculated as the Week 84 value minus the baseline value. Blood was drawn to analyze for CD4+ cell count.
Time Frame: Baseline and Week 84
Population: ITT-E Population, Randomized Phase. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 84 visit and had a cell count obtained during that visit period.
Measure: Mean (Standard Deviation); unit: cells/millimeters cubed (mm^3)
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 193 | 187
cells/millimeters cubed (mm^3) | 265.7 (157.65) | 282.9 (150.49)

17. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 144
Description: A CD4+ cell is a T lymphocyte that carries the CD4 antigen. Immunologic response was assessed by CD4+ counts. Change from baseline was calculated as the Week 144 value minus the baseline value. Blood was drawn to analyze for CD4+ cell count.
Time Frame: Baseline and Week 144
Population: ITT-Extension Population, Extension Phase. Observed Population. Participants withdrew as the study progressed; participants could only be included in the analysis if they had completed a Week 144 visit and had a cell count obtained during that visit period.
Measure: Mean (Standard Deviation); unit: cells/millimeters cubed (mm^3)
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 163 | 156
cells/millimeters cubed (mm^3) | 317.7 (161.98) | 325.1 (178.29)

18. Secondary Outcome: Number of Confirmed Virologic Failure Participants With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease From Baseline Through Week 36
Description: A blood sample was drawn for participants failing to respond to therapy, and the mutations present in the virus were identified. For each participant, the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New resistance-associated mutations (defined by the International AIDS Society-USA guidelines) that developed at the time of failure were tabulated by drug class. PAR, participants; VF, virologic failure; NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor.
Time Frame: Baseline through Week 36
Population: Participants in the ITT-E Population (Induction Phase) who met the confirmed virologic failure (CVF) criteria with paired baseline and virologic failure genotypic evaluations. One participant met CVF criteria at Week 36 and was randomized; these results are included in both the Week 36 and the Randomization through Week 84 results.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 15
participants
  PAR with paired genotypes at baseline and VF | 15
  PAR with treatment-emergent mutations | 6
  PAR with NRTI mutations | 4
  PAR with NNRTI mutations | 1
  PAR with major PI mutations | 0
  PAR with minor PI mutations | 2

19. Secondary Outcome: Number of Confirmed Virologic Failure Participants With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease From Randomization at Week 36 Through Week 84
Description: A blood sample was drawn for participants failing to respond to therapy, and the mutations present in the virus were identified. For each participant, the mutations found at the time of failure were compared with any mutations found in the blood sample at baseline. New International AIDs Society-USA defined resistance mutations that developed at the time of failure were tabulated by drug class. VF, virologic failure; NRTI, nucleoside reverse transcriptase inhibitor; NNRTI, non-nucleoside reverse transcriptase inhibitor; PI, protease inhibitor.
Time Frame: Randomization at Week 36 through Week 84
Population: Participants in the ITT-E Population (Randomized Phase) who met the confirmed virologic failure (CVF) criteria with paired baseline and virologic failure genotypic evaluations. One participant met CVF criteria at Week 36 and was randomized; these results are included in both the Week 36 and the Randomization through Week 84 results.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 1 | 7
participants
  PAR with paired genotypes at baseline and VF | 1 | 7
  PAR with treatment-emergent mutations | 1 | 2
  PAR with NRTI mutations | 1 | 0
  PAR with NNRTI mutations | 0 | 0
  PAR with major PI mutations | 0 | 0
  PAR with minor PI mutations | 0 | 2

20. Secondary Outcome: Number of Confirmed Virologic Failure Participants With Treatment-emergent HIV Genotypic Resistance in Reverse Transcriptase and Protease From Week 84 Through Week 144
Description: as for outcome 19
Time Frame: Week 84 through Week 144
Population: Participants in the ITT-Extension Population (Extension Phase) who met the confirmed virologic failure criteria with paired baseline and virologic failure genotypic evaluations.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 5 | 6
participants
  PAR with paired genotypes at baseline and VF | 5 | 5
  PAR with treatment-emergent mutations | 2 | 1
  PAR with NRTI mutations | 0 | 1
  PAR with NNRTI mutations | 0 | 0
  PAR with major PI mutations | 0 | 1
  PAR with minor PI mutations | 2 | 1

21. Secondary Outcome: Number of Confirmed Virologic Failure Participants From Baseline Through Week 36 With Treatment-emergent Reductions in Susceptibility to Abacavir, Lamivudine, Atazanavir, or Ritonavir
Description: A blood sample was drawn for participants failing to respond to therapy, and changes in drug susceptibility for HIV isolated from the participants for each drug used in the study were assessed. For each participant, the changes in drug susceptibility detected by phenotypic assay in virus from the sample collected at the time of failure was compared with drug susceptibility in the virus from the blood sample at baseline. PAR, participant.
Time Frame: Baseline through Week 36
Population: Participants in the ITT-E Population (Induction Phase) who met the confirmed virologic failure (CVF) criteria with paired baseline and virologic failure phenotypic evaluations. One participant met CVF criteria at Week 36 and was randomized; these results are included in both the Week 36 and the Randomization through Week 84 results.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 15
participants
  PAR with reduced abacavir susceptibility | 0
  PAR with reduced lamivudine susceptibility | 1
  PAR with reduced atazanavir susceptibility | 0
  PAR with reduced ritonavir susceptibility | 0

22. Secondary Outcome: Number of Confirmed Virologic Failure Participants From Randomization at Week 36 Through Week 84 With Treatment-emergent Reductions in HIV Susceptibility to Abacavir, Lamivudine, Atazanavir, or Ritonavir
Description: as for outcome 21
Time Frame: Randomization at Week 36 through Week 84
Population: Participants in the ITT-E population (Randomized Phase) who met the confirmed virologic failure (CVF) criteria with paired baseline and virologic failure phenotypic evaluations. One participant met CVF criteria at Week 36 and was randomized; these results are included in both the Week 36 and the Randomization through Week 84 results.
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 1 | 7
participants
  PAR with reduced abacavir susceptibility | 0 | 0
  PAR with reduced lamivudine susceptibility | 1 | 0
  PAR with reduced atazanavir susceptibility | 0 | 0
  PAR with reduced ritonavir susceptibility | 0 | 0

23. Secondary Outcome: Number of Confirmed Virologic Failure Participants From Week 84 Through Week 144 With Treatment-emergent Reductions in HIV Susceptibility to Abacavir, Lamivudine, Atazanavir, or Ritonavir
Description: as for outcome 21
Time Frame: Week 84 through Week 144
Population: Participants in the ITT-Extension Population (Extension Phase) who met the confirmed virologic failure criteria with paired baseline and virologic failure phenotypic evaluations
Measure: Number; unit: participants
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 5 | 6
participants
  PAR with reduced abacavir susceptibility | 0 | 1
  PAR with reduced lamivudine susceptibility | 1 | 1
  PAR with reduced atazanavir susceptibility | 0 | 1
  PAR with reduced ritonavir susceptibility | 0 | 1

24. Secondary Outcome: Mean Percent Compliance at Week 36
Description: Percent compliance is defined as the total number of pills taken divided by the total number of pills prescribed. The total number of pills taken was calculated by subtracting any returned pills from the total number of pills that were dispensed to each participant during this period. Compliance was calculated for each medication in the regimen.
Time Frame: Week 36
Population: ITT-E Population, Induction Phase. Participants with an unknown number of pills returned (including those whose pill bottles were not returned) were not included in this analysis.
Measure: Mean (Standard Deviation); unit: percent compliance
Arm/Group | ABC/3TC + ATV/r: Induction Phase
Number analyzed (Participants) | 503
percent compliance
  Abacavir/Lamivudine | 92.2 (13.05)
  Ritonavir | 92.3 (12.15)
  Atazanavir | 92.7 (12.50)

25. Secondary Outcome: Mean Percent Compliance at Week 84
Description: as for outcome 24
Time Frame: Week 84
Population: ITT-E Population, Randomized Phase. Participants with an unknown number of pills returned (including those whose pill bottles were not returned) were not included in this analysis.
Measure: Mean (Standard Deviation); unit: percent compliance
Arm/Group | ABC/3TC + ATV: Randomized Phase | ABC/3TC + ATV/r: Randomized Phase
Number analyzed (Participants) | 210 | 209
percent compliance
  Abacavir/Lamivudine | 92.0 (11.62) | 91.2 (13.49)
  Ritonavir | 92.9 (11.64) | 91.5 (12.23)
  Atazanavir | 98.9 (5.32) | 92.4 (11.89)

26. Secondary Outcome: Mean Percent Compliance at Week 144
Description: as for outcome 24
Time Frame: Week 144
Population: ITT-Extension Population, Extension Phase. Participants with an unknown number of pills returned (including those whose pill bottles were not returned) were not included in this analysis.
Measure: Mean (Standard Deviation); unit: percent compliance
Arm/Group | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Number analyzed (Participants) | 189 | 180
percent compliance
  Abacavir/Lamivudine | 92.0 (12.65) | 90.1 (15.35)
  Ritonavir | 93.3 (11.07) | 90.1 (14.58)
  Atazanavir | 99.1 (4.54) | 91.4 (13.99)

ADVERSE EVENTS:
Description: Data are cumulative. If an adverse event (AE) occurs in the Induction Phase (IP) at >=3%, and no new participants experience the AE in later phases, the participants who experienced the AE in the IP are carried over to the Randomization Phase and to the Extension Phase (if they remain in the study) if the incidence is >=3% for at least one arm.
Groups:
- ABC/3TC + ATV/r: Induction Phase: Induction Phase: participants in the Safety Population (participants exposed to at least one dose of investigational product) receiving abacavir (ABC) 600 milligrams (mg)/lamivudine (3TC) 300 mg fixed-dose combination tablet (FDC) once a day (QD) plus atazanavir (ATV) 300 mg QD + ritonavir (/r) 100 mg QD during the first 36 weeks of the study (planned interim analysis)
- ABC/3TC + ATV: Randomization Phase: Randomization Phase: participants in the Safety Population receiving a simplification regimen of the ABC/3TC FDC tablet administered QD for an additional 48 weeks in combination with ATV QD; includes serious adverse events (SAEs) that occurred during induction phase
- ABC/3TC + ATV/r: Randomization Phase: Randomization Phase: participants in the Safety Population receiving continuation of ABC/3TC FDC tablet administered QD for an additional 48 weeks in combination with ATV/r QD; includes SAEs that occurred during induction phase
- ABC/3TC + ATV: Extension Phase: Extension Phase: participants in the Safety Population receiving a simplification regimen of the ABC/3TC FDC tablet administered QD for an additional 60 weeks in combination with ATV QD
- ABC/3TC + ATV/r: Extension Phase: participants in the Safety Population receiving continuation of ABC/3TC FDC tablet administered QD for an additional 60 weeks in combination with ATV/r QD
Arm/Group | ABC/3TC + ATV/r: Induction Phase | ABC/3TC + ATV: Randomization Phase | ABC/3TC + ATV/r: Randomization Phase | ABC/3TC + ATV: Extension Phase | ABC/3TC + ATV/r: Extension Phase
Serious Adverse Events (participants affected / at risk) | 39/515 | 22/210 | 22/209 | 24/189 | 24/180
Other Adverse Events (participants affected / at risk) | 237/515 | 116/210 | 123/209 | 123/189 | 130/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABC/3TC + ATV/r: Induction Phase (N=515) | ABC/3TC + ATV: Randomization Phase (N=210) | ABC/3TC + ATV/r: Randomization Phase (N=209) | ABC/3TC + ATV: Extension Phase (N=189) | ABC/3TC + ATV/r: Extension Phase (N=180)
Appendicitis (Infections and infestations) | 3 | 2 | 1 | 1 | 2
Appendicitis, perforated (Infections and infestations) | 0 | 1 | 1 | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 2 | 0
Cellulitis (Infections and infestations) | 1 | 2 | 0 | 4 | 0
Peritoneal infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Shigella infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Proctitis gonococcal (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 5 | 2 | 3 | 1 | 4
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 2 | 1 | 1 | 1 | 0
Syncope (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2 | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 1
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Burkitt's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Pharyngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1
Mental disorder (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 0 | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABC/3TC + ATV/r: Induction Phase (N=515) | ABC/3TC + ATV: Randomization Phase (N=210) | ABC/3TC + ATV/r: Randomization Phase (N=209) | ABC/3TC + ATV: Extension Phase (N=189) | ABC/3TC + ATV/r: Extension Phase (N=180)
Diarrhoea (Gastrointestinal disorders) | 42 | 24 | 23 | 25 | 21
Blood bilirubin increased (Hepatobiliary disorders) | 40 | 20 | 22 | 22 | 24
Hyperbilirubinaemia (Hepatobiliary disorders) | 30 | 14 | 20 | 14 | 20
Nausea (Gastrointestinal disorders) | 24 | 12 | 10 | 9 | 12
Rash (Skin and subcutaneous tissue disorders) | 23 | 10 | 7 | 10 | 7
Sinusitis (Infections and infestations) | 21 | 15 | 19 | 19 | 25
Bronchitis (Infections and infestations) | 18 | 11 | 22 | 20 | 22
Depression (Psychiatric disorders) | 18 | 11 | 10 | 11 | 15
Insomnia (Psychiatric disorders) | 17 | 6 | 11 | 11 | 13
Headache (Nervous system disorders) | 16 | 10 | 10 | 9 | 9
Upper respiratory tract infection (Infections and infestations) | 16 | 13 | 16 | 20 | 19
Anxiety (Psychiatric disorders) | 12 | 9 | 8 | 10 | 7
Blood Cholesterol increased (Investigations) | 8 | 7 | 7 | 8 | 7
Fatigue (General disorders) | 4 | 5 | 8 | 6 | 8
Syphilis (Infections and infestations) | 7 | 5 | 7 | 12 | 10
Lipase increased (Investigations) | 4 | 8 | 1 | 9 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 7 | 0 | 11 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 3 | 3 | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 3 | 8 | 5
Blood triglycerides increased (Investigations) | 8 | 4 | 4 | 6 | 6
Cellulitis (Infections and infestations) | 5 | 6 | 3 | 9 | 3
Influenza (Infections and infestations) | 9 | 6 | 4 | 6 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 4 | 4 | 3 | 8
Abdominal pain (Gastrointestinal disorders) | 4 | 6 | 3 | 6 | 4
Hypertension (Vascular disorders) | 1 | 1 | 4 | 2 | 8
Nasopharyngitis (Infections and infestations) | 7 | 2 | 6 | 2 | 8
Conjunctivitis (Eye disorders) | 7 | 3 | 4 | 3 | 6
Vomiting (Gastrointestinal disorders) | 9 | 6 | 4 | 6 | 3
Low density lipoprotein increased (Investigations) | 4 | 4 | 3 | 6 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 6 | 5 | 1 | 6 | 1
Pneumonia (Infections and infestations) | 4 | 0 | 4 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.